CLINICAL TRIAL: NCT02958293
Title: Does Procedural Timing Impact Perioperative Morbidity in Elective Surgery?
Brief Title: Perioperative Morbidity in Elective Surgery Based on the Time of the Year
Status: Completed | Type: Observational
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 16-049
Record Dates: First submitted 2016-11-02; First posted 2016-11-08 (Estimated); Results first posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2022-10

CONDITIONS: Perioperative Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a retrospective cohort study using Electronic Privacy Identification Center (EPIC) database to evaluate if there are any differences in perioperative morbidity for elective surgery based on the time of the year surgery is performed.

DETAILED DESCRIPTION:
Surgical complications are a significant cause of morbidity and mortality. Surgical complications account for up to 40% of hospital complications. Complications and adverse events are also becoming increasingly important for measuring health care quality.

Many physician practices notice a surge of patients seeking care at the end of the year compared to other times of the year. Patients who meet their insurance deductibles are likely more eager to proceed with an elective procedure. Patients who have met their deductible likely utilize more healthcare resources because they have more health problems, or have had more procedures performed during that year. Thus there may be potential for sicker and more complicated patients to undergo surgery at the end of the year as compared to other times of the year.

Prior studies have often evaluated the "July effect" which is the beginning of a new academic year at teaching hospitals. Not only are new interns involved in patient care but trainees at all levels are in participating in a new role. Several prior studies have found high morbidity and mortality rates in July-August compared to April-June. There is paucity of research evaluating the measures for the months of November-December.

Identifying which patients are at a higher risk for perioperative morbidity is important to help prevent surgical complications and lower healthcare costs. Proper patient selection and appropriate timing for elective procedures will positively impact these adverse outcomes.

This study is a retrospective cohort study investigating whether there are differences in perioperative morbidity for elective surgery based on the time of the year surgery is performed. The results of this project could impact counseling for patient regarding timing of their surgery based on calendar month. This could also help implement changes in how systems based care is provided regarding insurance deductibles and maximums.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 and older undergoing surgical procedures in the main operating room between July 1, 2012 and July 1, 2016.

Exclusion Criteria:

* Patients under the age of 18
* Procedures done outside of the main operating suites (Endoscopy suite, Labor and Delivery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent a surgical procedure in the main operating rooms at Good Samaritan Hospital and Bethesda North Hospital
Sampling Method: Non-Probability Sample
Enrollment: 19872 (Actual)
Dates: Start 2016-11; Primary Completion 2018-03-26 (Actual); Study Completion 2018-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Pauls, MD, Principal Investigator — TriHealth - Cincinnati Urogynecology Associates

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Surgery: All patients 18 years and older who underwent a surgical procedure in the main operating rooms at Good Samaritan Hospital and Bethesda North Hospital between January 1, 2015 and December 31, 2016.
  Equal numbers of charts were randomly selected for each calendar month.
Period: Overall Study
Arm/Group | Patients With Surgery
Started | 19872
Completed | 19872
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Patients With Surgery: All patients 18 years and older who underwent a surgical procedure in the main operating rooms at Good Samaritan Hospital and Bethesda North Hospital between January 1, 2015 and December 31, 2016.
Arm/Group | Patients With Surgery
Number analyzed (Participants) | 19872
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.68 (16.13)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 12448
  Male | 7423
  Unknown | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 16726
  African American | 2403
  Other | 743
Region of Enrollment [Number; unit: participants]
  United States | 19872

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Surgical Complication
Description: All patients 18 years and older who underwent a surgical procedure in the main operating rooms at Good Samaritan Hospital and Bethesda North Hospital between January 1, 2015 and December 31, 2016.
Time Frame: 90 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Surgery
Number analyzed (Participants) | 19872
Participants | 3513

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Patients With Surgery
All-Cause Mortality (participants affected / at risk) | 0/19872
Serious Adverse Events (participants affected / at risk) | 0/19872
Other Adverse Events (participants affected / at risk) | 0/19872

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-09): https://cdn.clinicaltrials.gov/large-docs/93/NCT02958293/Prot_SAP_000.pdf